CLINICAL TRIAL: NCT05465226
Title: A pRospective, Case-controlled Evaluation of oLIceridine for Moderate or sEVEre Pain in Patients With Acute Burn Injuries. (RELIEVE)
Brief Title: Oliceridine in Patients With Acute Burn Injuries
Acronym: RELIEVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-08748-FB
Record Dates: First submitted 2022-06-22; First posted 2022-07-19 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Pain; Burns; Adverse Drug Event; Respiratory Depression; Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Acute Pain; Burns; Drug-Related Side Effects and Adverse Reactions; Respiratory Insufficiency; Postoperative Nausea and Vomiting | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, prospective, case-controlled trial. Intervention arm patients will be randomly matched 2:1 to a historical comparator, based on age, TBSA, number of surgeries, and opioid and illicit drug use histories
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oliceridine Arm (Experimental): Initially, patients will receive oliceridine 1-3 mg IVP every 1-3 hours as needed for moderate or severe pain (NRS ≥ 4) with 1-3 mg every 1-3 hours for breakthrough pain. NRS will be assessed every 3-4 hours routinely. Rescue doses will be allowed per clinical discretion as oliceridine 1-3 mg every hour. Doses will be titrated according to patient response and clinical discretion. In settings where rapid analgesia is needed, such as the operating room, post-anesthesia care unit, emergency room, or hydrotherapy, oliceridine will be administered in 0.5-2 mg doses every 5 minutes as needed for moderate or severe pain, according to anesthesiologist or treating physician's discretion. For the purposes of the study oliceridine will not exceed 7 days of administration and patients will be transitioned from intravenous opioids to oral therapy and de-escalated from opioids, as soon as the team deems appropriate.
  Interventions: Drug: Oliceridine
- Historical control (Active Comparator): Retrospective, observational, historical control arm matched by age, TBSA, number of surgeries, and opioid and illicit drug use histories
  Interventions: Drug: Historical opioid use

INTERVENTIONS:
Drug: Oliceridine — see arm description
  Arms: Oliceridine Arm
Drug: Historical opioid use — Historical matched, control group in 2:1 ratio
  Arms: Historical control

SUMMARY:
Pain after acute burn injury is complex with much still not understood. The primary mechanism is believed to be nociceptive, but is interwoven with aspects of somatogenic, neuropathic, and psychogenic pathways. As such, opioid receptor agonists are an essential component for pain management after burn injury. The majority of wound care and dressing changes are completed in non-intubated patients and rates of respiratory depression concerning. Oliceridine is a biased, selective MOR agonist approved for treatment of acute pain. To date there is no literature of use in patients with burn injuries. While it should be effective, efficacy and the potential for reduced adverse events need to be quantified. Current practice and guidelines, plead for better analgesia for patients with burn injuries.

DETAILED DESCRIPTION:
Pain after acute burn injury is complex with much still not understood. After acute burn injury, both injured tissue and adjacent non-burned tissue, upregulate response to painful and non-painful stimulus (hyperalgesia and allodynia, respectively). The primary mechanism is believed to be nociceptive, but is interwoven with aspects of somatogenic, neuropathic, and psychogenic pathways. As such, opioid receptor agonists are an essential component for pain management after burn injury. Currently, high-dose fentanyl, oxycodone, hydromorphone, and morphine are used at profound doses to mitigate pain associated with daily care of patients with burn injuries. The majority of wound care and dressing changes are completed in non-intubated patients and rates of respiratory depression concerning.

High-quality data is controversial or lacking on the best approach for multimodal analgesia. Additionally, limitations exist for prescribing and monitoring some agents. While a multimodal approach may lead to a reduction in acute or chronic pain, adding a handful of medicines to eliminate a single agent leads to exponentially more side effects, risk of adverse effects, drug interactions, and pill burden. Drugs targeting neuropathic pain delay neural processing and are accompanied by cognitive slowing and responsiveness, which increases fall risk and limits rehabilitation participation. Gabapentin and pregabalin efficacies are highly debated with variable dosing recommendations. Side effects are common and include dizziness, somnolence, confusion, vision loss, respiratory dysfunction, peripheral edema, gastrointestinal discomfort or irregularities, or asthenia. If effective, serotonin-norepinephrine reuptake inhibitors response can be delayed by weeks and are known to cause significant weight loss, dizziness, asthenia, sleep disorders, and gastrointestinal dysfunction. Acetaminophen can help reduce background pain, but is hepatotoxic, depletes glutathione, and can mask fever. Nonsteroidal anti-inflammatory drugs carry significant safety concerns, including cardiovascular events, platelet dysfunction, bleeding, gastrointestinal toxicity, and renal failure. Local anesthetics have limited efficacy and dissipate quickly. Peripheral nerve blocks have mostly been studied for donor site pain, and placement requires specialized skills. Ketamine can be extremely helpful, especially in non-naïve patients with high-opioid tolerances but is approved as a moderate sedative and many state laws limit who can prescribe and/or monitor its administration. While ketamine does not depress respiratory drive, it is a hallucinogen, pro-deliriogenic, pro-arrhythmogenic, and carries its own concerns for gastrointestinal irregularities and drug dependence.

Opioid agonists bind to the mu opioid receptor (MOR), triggering downstream signaling through either G-protein-coupled or β-arrestin pathways. While the G-protein pathway is primarily involved in analgesia, β-arrestin has been shown responsible for adverse events, especially respiratory depression and gastrointestinal dysfunction. Additionally, the β-arrestin pathway terminates G-protein activation and induces endocytosis of the receptor, which can lead to reduced analgesia or opioid tolerance. Oliceridine is a biased, selective MOR agonist approved for treatment of acute pain. Oliceridine has shown a 3-fold preferential pathway activation of G-protein over β-arrestin. As a result, subsequent clinical trials have resulted in improved analgesia over placebo and morphine, while significantly reducing adverse events. To date there is no literature of use in patients with burn injuries. While it should be effective, efficacy and the potential for reduced adverse events need to be quantified. Current practice and guidelines, plead for better analgesia for patients with burn injuries.

ELIGIBILITY:
Inclusion Criteria:

* 1) age ≥ 18 years old,
* 2) total body surface area (TBSA) burned < 20%
* 3) deep partial thickness or full thickness burns admitted for possible or definitive surgical needs,
* 4) moderate or severe pain related to acute burns (NRS ≥ 4 out of 10)

Exclusion Criteria:

* 1) Presence of inhalation injury,
* 2) Pregnant,
* 3) Incarcerated,
* 4) only initial admission,
* 5) known anaphylaxis to oliceridine or other opioids,
* 6) Patient or authorized representative unable or unwilling to consent,
* 7) known cocaine, methamphetamine, or opioid use history,
* 8) use of numeric rating scale (NRS) would be inaccurate or inappropriate
* 9) Significant hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Analyze change in pain scores after initiation of oliceridine in patients with moderate or severe pain after acute burn injury | Baseline and every 3-4 hours as standard of care allows or study medication continued, up to 7 days
  Change in Numeric Rating Scale (0 - 10 with 10 being the worst) pain scores after initiation

SECONDARY OUTCOMES:
Characterize adverse events associated with administration of oliceridine in patients with acute burn injury | At least daily while taking study medication, up to 7 days
  Monitor for adverse events
Establish a burn injury-specific half maximal effective concentration | Sparse sampling strategy with up to 6 samples taken over the 4-hour dosing scheme
  Plasma samples to measure concentration and pair with numeric pain score captured for Outcome 1
Establish a burn injury-specific half-life | Sparse sampling strategy with up to 6 samples taken over the 4-hour dosing scheme
  Plasma samples to measure concentrations and calculate elimination coefficient
Establish a burn injury-specific volume of distribution | Sparse sampling strategy with up to 6 samples taken over the 4-hour dosing scheme
  Plasma samples to measure concentrations and calculate volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James DL, Jowza M. Principles of Burn Pain Management. Clin Plast Surg. 2017 Oct;44(4):737-747. doi: 10.1016/j.cps.2017.05.005. Epub 2017 Jul 15. PMID 28888299
- [Background] Romanowski KS, Carson J, Pape K, Bernal E, Sharar S, Wiechman S, Carter D, Liu YM, Nitzschke S, Bhalla P, Litt J, Przkora R, Friedman B, Popiak S, Jeng J, Ryan CM, Joe V. American Burn Association Guidelines on the Management of Acute Pain in the Adult Burn Patient: A Review of the Literature, a Compilation of Expert Opinion and Next Steps. J Burn Care Res. 2020 Nov 30;41(6):1152-1164. doi: 10.1093/jbcr/iraa120. No abstract available. PMID 32885252
- [Background] Thompson EM, Andrews DD, Christ-Libertin C. Efficacy and safety of procedural sedation and analgesia for burn wound care. J Burn Care Res. 2012 Jul-Aug;33(4):504-9. doi: 10.1097/BCR.0b013e318236fe4f. PMID 22079919
- [Background] Myers R, Lozenski J, Wyatt M, Pena M, Northrop K, Bhavsar D, Kovac A. Sedation and Analgesia for Dressing Change: A Survey of American Burn Association Burn Centers. J Burn Care Res. 2017 Jan/Feb;38(1):e48-e54. doi: 10.1097/BCR.0000000000000423. PMID 27606558
- [Background] Wibbenmeyer L, Oltrogge K, Kluesner K, Zimmerman MB, Kealey PG. An evaluation of discharge opioid prescribing practices in a burn population. J Burn Care Res. 2015 Mar-Apr;36(2):329-35. doi: 10.1097/BCR.0000000000000110. PMID 25680091
- [Background] Wibbenmeyer L, Eid A, Kluesner K, Heard J, Zimmerman B, Kealey GP, Brennan T. An Evaluation of Factors Related to Postoperative Pain Control in Burn Patients. J Burn Care Res. 2015 Sep-Oct;36(5):580-6. doi: 10.1097/BCR.0000000000000199. PMID 26335109
- [Background] Kaul I, Amin A, Rosenberg M, Rosenberg L, Meyer WJ 3rd. Use of gabapentin and pregabalin for pruritus and neuropathic pain associated with major burn injury: A retrospective chart review. Burns. 2018 Mar;44(2):414-422. doi: 10.1016/j.burns.2017.07.018. Epub 2017 Aug 16. PMID 28822592
- [Background] Wibbenmeyer L, Eid A, Liao J, Heard J, Horsfield A, Kral L, Kealey P, Rosenquist R. Gabapentin is ineffective as an analgesic adjunct in the immediate postburn period. J Burn Care Res. 2014 Mar-Apr;35(2):136-42. doi: 10.1097/BCR.0b013e31828a4828. PMID 23511293
- [Background] Jones LM, Uribe AA, Coffey R, Puente EG, Abdel-Rasoul M, Murphy CV, Bergese SD. Pregabalin in the reduction of pain and opioid consumption after burn injuries: A preliminary, randomized, double-blind, placebo-controlled study. Medicine (Baltimore). 2019 May;98(18):e15343. doi: 10.1097/MD.0000000000015343. PMID 31045775
- [Background] Meyer WJ 3rd, Nichols RJ, Cortiella J, Villarreal C, Marvin JA, Blakeney PE, Herndon DN. Acetaminophen in the management of background pain in children post-burn. J Pain Symptom Manage. 1997 Jan;13(1):50-5. doi: 10.1016/s0885-3924(96)00201-1. PMID 9029861
- [Background] Retrouvey H, Shahrokhi S. Pain and the thermally injured patient-a review of current therapies. J Burn Care Res. 2015 Mar-Apr;36(2):315-23. doi: 10.1097/BCR.0000000000000073. PMID 24823343
- [Background] Pal SK, Cortiella J, Herndon D. Adjunctive methods of pain control in burns. Burns. 1997 Aug;23(5):404-12. doi: 10.1016/s0305-4179(97)00029-6. PMID 9426910
- [Background] Yang C, Xu XM, He GZ. Efficacy and feasibility of opioids for burn analgesia: An evidence-based qualitative review of randomized controlled trials. Burns. 2018 Mar;44(2):241-248. doi: 10.1016/j.burns.2017.10.012. Epub 2017 Nov 21. PMID 29169696
- [Background] Ly E, Velamuri S, Hickerson W, Hill DM, Desai J, Tsui B, Herr M, Jones J. Approaching trauma analgesia using prolonged and novel continuous peripheral nerve blocks - A case report. Anesth Pain Med (Seoul). 2022 Jan;17(1):87-92. doi: 10.17085/apm.21029. Epub 2021 Jul 22. PMID 34784461
- [Background] MacPherson RD, Woods D, Penfold J. Ketamine and midazolam delivered by patient-controlled analgesia in relieving pain associated with burns dressings. Clin J Pain. 2008 Sep;24(7):568-71. doi: 10.1097/AJP.0b013e31816cdb20. PMID 18716494
- [Background] Lintner AC, Brennan P, Miles MVP, Leonard C, Alexander KM, Kahn SA. Oral Administration of Injectable Ketamine During Burn Wound Dressing Changes. J Pharm Pract. 2021 Jun;34(3):423-427. doi: 10.1177/0897190019876497. Epub 2019 Sep 19. PMID 31537149
- [Background] Brennan PG, Landry JK, Miles MVP, Lintner AC, McGinn KA, Kahn SA. Intravenous Ketamine as an Adjunct to Procedural Sedation During Burn Wound Care and Dressing Changes. J Burn Care Res. 2019 Feb 20;40(2):246-250. doi: 10.1093/jbcr/iry044. PMID 30189001
- [Background] DeWire SM, Ahn S, Lefkowitz RJ, Shenoy SK. Beta-arrestins and cell signaling. Annu Rev Physiol. 2007;69:483-510. doi: 10.1146/annurev.physiol.69.022405.154749. PMID 17305471
- [Background] Raehal KM, Walker JK, Bohn LM. Morphine side effects in beta-arrestin 2 knockout mice. J Pharmacol Exp Ther. 2005 Sep;314(3):1195-201. doi: 10.1124/jpet.105.087254. Epub 2005 May 25. PMID 15917400
- [Background] Luttrell LM, Lefkowitz RJ. The role of beta-arrestins in the termination and transduction of G-protein-coupled receptor signals. J Cell Sci. 2002 Feb 1;115(Pt 3):455-65. doi: 10.1242/jcs.115.3.455. PMID 11861753
- [Background] DeWire SM, Yamashita DS, Rominger DH, Liu G, Cowan CL, Graczyk TM, Chen XT, Pitis PM, Gotchev D, Yuan C, Koblish M, Lark MW, Violin JD. A G protein-biased ligand at the mu-opioid receptor is potently analgesic with reduced gastrointestinal and respiratory dysfunction compared with morphine. J Pharmacol Exp Ther. 2013 Mar;344(3):708-17. doi: 10.1124/jpet.112.201616. Epub 2013 Jan 8. PMID 23300227
- [Background] Viscusi ER, Skobieranda F, Soergel DG, Cook E, Burt DA, Singla N. APOLLO-1: a randomized placebo and active-controlled phase III study investigating oliceridine (TRV130), a G protein-biased ligand at the micro-opioid receptor, for management of moderate-to-severe acute pain following bunionectomy. J Pain Res. 2019 Mar 11;12:927-943. doi: 10.2147/JPR.S171013. eCollection 2019. PMID 30881102
- [Background] Singla NK, Skobieranda F, Soergel DG, Salamea M, Burt DA, Demitrack MA, Viscusi ER. APOLLO-2: A Randomized, Placebo and Active-Controlled Phase III Study Investigating Oliceridine (TRV130), a G Protein-Biased Ligand at the mu-Opioid Receptor, for Management of Moderate to Severe Acute Pain Following Abdominoplasty. Pain Pract. 2019 Sep;19(7):715-731. doi: 10.1111/papr.12801. Epub 2019 Jun 24. PMID 31162798
- [Background] Bergese SD, Brzezinski M, Hammer GB, Beard TL, Pan PH, Mace SE, Berkowitz RD, Cochrane K, Wase L, Minkowitz HS, Habib AS. ATHENA: A Phase 3, Open-Label Study Of The Safety And Effectiveness Of Oliceridine (TRV130), A G-Protein Selective Agonist At The micro-Opioid Receptor, In Patients With Moderate To Severe Acute Pain Requiring Parenteral Opioid Therapy. J Pain Res. 2019 Nov 14;12:3113-3126. doi: 10.2147/JPR.S217563. eCollection 2019. PMID 31814753
- [Background] Nafziger AN, Arscott KA, Cochrane K, Skobieranda F, Burt DA, Fossler MJ. The Influence of Renal or Hepatic Impairment on the Pharmacokinetics, Safety, and Tolerability of Oliceridine. Clin Pharmacol Drug Dev. 2020 Jul;9(5):639-650. doi: 10.1002/cpdd.750. Epub 2019 Nov 7. PMID 31697049
- [Background] Fossler MJ, Sadler BM, Farrell C, Burt DA, Pitsiu M, Skobieranda F, Soergel DG. Oliceridine (TRV130), a Novel G Protein-Biased Ligand at the mu-Opioid Receptor, Demonstrates a Predictable Relationship Between Plasma Concentrations and Pain Relief. I: Development of a Pharmacokinetic/Pharmacodynamic Model. J Clin Pharmacol. 2018 Jun;58(6):750-761. doi: 10.1002/jcph.1076. Epub 2018 Feb 7. PMID 29412458